CLINICAL TRIAL: NCT01821638
Title: Brain Alterations and Cognitive Impairment in Older Adults With Heart Failure
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2012-1064
Record Dates: First submitted 2013-03-20; First posted 2013-04-01 (Estimated); Last update posted 2019-02-06 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure
Keywords: Heart failure; Cognition; Brain; Older adults
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Older adults with heart failure: Older adults with heart failure

SUMMARY:
Cognitive impairment, commonly reported as difficulty with memory and executive function, is a widely recognized clinical challenge for older persons with heart failure (HF). Little is known about the relationship between brain MRI and cognitive impairment in older persons with HF. A limited number of studies have investigated brain MRI in adults with HF and produced conflicting results. Previous findings are limited by use of lower resolution scanners (1.5 Tesla), lack of MRI techniques (i.e. combining structural sequences with perfusion sequences) and recruitment of mixed age samples. Based on these limitations, the purpose of this research plan is to explore the relationship between brain MRI and cognitive impairment in older persons with HF using high resolution structural and perfusion scans. To accomplish this goal, investigators will compare 40 adults with HF who are age > 65 years old with 40 healthy, gender, age, and education matched controls. Investigators will obtain neuropsychological measures of multiple domains, as well as MRI measurements of the temporal lobe and prefrontal cortex at baseline and 12-months.

DETAILED DESCRIPTION:
Cognitive impairment, commonly reported as difficulty with memory and executive function, is a widely recognized clinical challenge for persons > 65 years old with HF. Although the degree of cognitive impairment usually does not meet the criteria for dementia, it can affect an individual's ability to process and remember information, such as complex medication regimens [5]. Findings suggest that brain regions that support memory (i.e. temporal lobe) and executive function (i.e. prefrontal cortex) may be altered in older persons with HF; suggesting that these brain alterations are related to the HF disease process and not normal aging. Surprisingly, despite the high prevalence of cognitive impairment in HF, relationships between brain and cognition have not been well studied.

Little is known about the relationships between brain magnetic resonance imaging (MRI) and cognitive impairment in older persons with HF. A limited number of studies have investigated brain MRI in adults with HF and produced conflicting results. Three studies utilized structural MRI techniques and identified evidence of atrophy in the temporal lobe, hippocampus, and prefrontal cortex and an increased volume of white matter hyperintensities [6-8]. Brain hypoperfusion, operationalized as decreased global cerebral perfusion, was identified in two studies [9, 10]. Only one study examined relationships between brain MRI and cognitive impairment in HF [6]. Vogels et al., (2007) found that atrophy in the medial temporal lobe was associated with decreased measures of memory and executive function. White matter hyperintensities did not correlate with any cognitive measures. Limited research findings indicate that various brain alterations in the temporal lobe, hippocampus, and prefrontal cortex contribute to cognitive impairment in HF. However, previous findings are limited by use of lower resolution scanners (1.5 Tesla), lack of MRI techniques (i.e. structural and perfusion scans) and recruitment of mixed age samples.

Based on these limitations, the purpose of this research plan is to explore relationships between brain MRI and cognitive impairment in older persons with HF using high resolution structural and perfusion scans. To accomplish this goal, investigators will compare 40 adults with HF who are > 65 years old with 40 healthy, gender, age, and education matched controls. Investigators will obtain neuropsychological measures of multiple domains, as well as MRI measurements of the temporal lobe and prefrontal cortex at baseline and 12-months. The following specific aims will be investigated:

Aim 1: Compare brain MRI in older persons with HF and controls at baseline and 12-months.

Hypothesis 1a: Older persons with HF will have increased white matter hyperintensities, decreased grey matter volume, and decreased perfusion in the temporal lobe and prefrontal cortex compared with controls. Hypothesis 1b: Older persons with HF will exhibit a greater decline in grey matter volume in the temporal lobe and prefrontal cortex over 12-months compared with controls.

Aim 2: Compare cognitive function in older persons with HF and controls at baseline and 12-months.

Hypothesis 2a): Older persons with HF will perform lower on measures of memory and executive function compared with controls.

Hypothesis 2b): Older persons with HF will exhibit a greater decline on measures of memory and executive function over 12-months compared with controls.

Aim 3: Examine the relationships between brain MRI and cognitive function in older persons with HF and controls at baseline.

Hypothesis 3a: Decreased grey matter and perfusion in the temporal lobe and an increased volume of white matter hyperintensities in the temporal lobe will be associated with decreased memory scores.

Hypothesis 3b: Decreased grey matter and perfusion in the prefrontal cortex and an increased volume of white matter hyperintensities in the prefrontal cortex will be associated with a decreased executive function score.

ELIGIBILITY:
Inclusion Criteria:

* 65 years old or older
* English speaking and writing;
* Stable guideline based medication regimen for at least four weeks prior to enrollment
* New York Heart Association classification I-IV

Exclusion Criteria:

* Mini-Mental Status Exam score equal to or less than 24;
* Current diagnosis of neurological illnesses or movement disorders (e.g. Alzheimer's dementia, Parkinson's disease, Epilepsy);
* History of substance abuse/treatment;
* Untreated depression
* History of stroke;
* Hepatic insufficiency;
* Severe renal failure;
* Untreated anemia;
* Left ventricular assist device;
* History of the following within three months of study enrollment: acute myocardial infarction, unstable angina, coronary artery bypass surgery, percutaneous transluminal angioplasty, or biventricular pacemaker insertion;
* History of implantable device (or other MRI contraindications).
* Prisoners
* Pregnancy

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Older adults with heart failure
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Mean neuropsychological test scores and brain changes | One year
  Compare mean values of the following outcomes between older adults with heart failure and older adults without heart failure at baseline
  * neuropsychological test scores
  * brain medial temporal lobe volume
  * brain frontal cortex volume
  * brain medial temporal lobe perfusion
  * brain frontal cortex perfusion
  Compare mean value changes in the following outcomes between baseline and one year in patients with heart failure:
  * neuropsychological test scores
  * brain medial temporal lobe volume
  * brain frontal cortex volume
  * brain medial temporal lobe perfusion
  * brain frontal cortex perfusion

CONTACTS AND LOCATIONS:
Overall Officials: Lisa C Bratzke, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No